CLINICAL TRIAL: NCT03640169
Title: Evaluation Project for the Development of Health Management Model for Chinese Medical Preventive Medicine
Brief Title: Development of Health Management Model for Chinese Medical Preventive Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, China (Other); Tri-Service General Hospital (Other); Taiwan Society of Health Promotion (Unknown); National Research Institute of Chinese Medicine, Ministry of Health and Welfare (Other Government); National Yang Ming Chiao Tung University (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yi-Chang Su, Professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMUH106-REC1-082
Record Dates: First submitted 2018-07-20; First posted 2018-08-21 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Preventive Medicine; Health Promotion
Keywords: Health Management Model; Chinese Medicine; Preventive Medicine; Body Constitution; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Management of TCM preventive medicine (Experimental): The Health management model include: (1) Body constitution measurement (2) Health promotion literacy education lectures (3) Duo-in qigong practice.
  Interventions: Other: Health management of TCM preventive medicine

INTERVENTIONS:
Other: Health management of TCM preventive medicine — The Health management model include: (1) Body constitution measurement (2) Health promotion literacy education lectures (3) Duo-in qigong practice.

SUMMARY:
The purpose of this project is to design a health management model of TCM preventive medicine that meets the need of healthy or suboptimal healthy people. This project will try to practice "Health management model of TCM preventive medicine" together with health promotion groups related to Taiwan Society of Health Promotion in the district of Shilin and Zhongzheng in Taipei city, and plan to recruit 100 people.

DETAILED DESCRIPTION:
With regard to "Developing traditional Chinese medicine (TCM) Health Care", the goal of "Promoting the development of TCM health promotion service" was set and the strategy of "Promoting the development of TCM preventive medicine and health promotion services" was used to develop TCM preventive medicine, which is applied to preventing disease and improving physical fitness. By establishing the TCM health care prototype of "health promotion" and "preventive medicine," this project will push the systemic development of TCM preventive medicine forward and improve suboptimal health by early intervention, providing people with multiple model choices in self-health management.

This project will first form a multidisciplinary team to gather and analyze the domestic and international health promotion and management models of TCM or traditional medicine. Then systematically arrange and induct the literature references to establish the outline and draft of "Health management model of TCM preventive medicine." Furthermore, in July-September, this project will try to practice "Health management model of TCM preventive medicine" together with health promotion groups related to Taiwan Society of Health Promotion in the district of Shilin and Zhongzheng in Taipei city, and plan to recruit 100 people. The purpose of this project is to design a health management model of TCM preventive medicine that meets the need of healthy or suboptimal healthy people. The investigators expecte to bring out the prototype of "Health management model of TCM preventive medicine" and finish the follow-up promoting proposal of the draft in the meantime, which will discuss the possibility of applying this model to healthy or suboptimal healthy people and bring up concrete policy and implementation recommendations of "promoting the development of TCM preventive medicine and health promotion services."

ELIGIBILITY:
Inclusion Criteria:

* more than 20 y/o.
* can walk independently, without disability
* can communicate with Chinese or Taiwanese, and understand the purpose of the study

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2017-09-16 (Actual)

PRIMARY OUTCOMES:
Body Constitution Scores (measured by Body Constitution Questionnaire, BCQ) | Change from Baseline Body Constitution Yang- deficiency, Yin- deficiency and Stasis Scores at 8 week
  The measurement of Body Constitution Questionnaire will come out 3 scores:
  Scores of Yang-deficiency: ranged from 19-95 Score of Yin- deficiency: ranged from 19-95 Score of Stasis: ranged from 16-80 The higher the score, the worse the Yang- deficiency, Yin- deficiency and Stasis.
Blood pressure | Change from baseline of both systolic and diastolic pressure at 8 week
  Change of both systolic and diastolic pressure after 8 week
Heart rate | Change from Baseline Heart rate at 8 week
  Change of Heart rate after 8 week
Heart rate variability | Change from Baseline Heart rate variability at 8 week
  Change of Heart rate variability after 8 week
Blood oxygen concentration | Change from Baseline Blood oxygen concentration at 8 week
  Change of Blood oxygen concentration after 8 week
Pittsburgh Sleep Quality Index | Change from Baseline total score of Pittsburgh Sleep Quality Index at 8 week
  Change of the global score of Pittsburgh Sleep Quality Index after 8 week The higher the global score, the worse the sleep quality. If the global <=5, defined to have good sleep quality; If the global > 5, defined to have bad sleep quality.
Brief Symptom Rating Scale（BSRS-5） | Change from Baseline BSRS-5 at 8 week
  Change of the score of the Brief Symptom Rating Scale after 8 week. Score ranged from 0-24: the higher the score the worse the physical and mental condition.
Dietary behavior Instrument | Change from Baseline total score of the Dietary behavior Instrument at 8 week
  Change of score of the Dietary behavior Instrument after 8 week. Score ranged from 0-36: the higher the score, the better the eating behavior.
Pressure index | Change from Baseline score of Pressure index at 8 week
  Change of the pressure feeling after 8 week. Score ranged from 0-12: the higher the score, the heavy the pressure feeling.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chang Su, PhD, Principal Investigator — China Medical University, China
Locations (1):
- Taiwan Society of Health Promotion, Taipei, Taiwan

REFERENCES:
- [Derived] Tsai YN, Chang YH, Su YC, Lee SM, Hsiao CH, Lin CK, Lin SJ. A community-based Daoyin program for health promotion: effects of the Qi and mind harmonizing method on body constitution for the health of older adults. Front Public Health. 2026 Jan 5;13:1644273. doi: 10.3389/fpubh.2025.1644273. eCollection 2025. PMID 41561842